CLINICAL TRIAL: NCT05906680
Title: The Gut Virome as a Trigger for IBD: From Metagenomics to Pathogenesis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Silvio Danese, Gastroenterologist, IRCCS San Raffaele
Other Study IDs: IBDomic
Record Dates: First submitted 2023-06-07; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: IBD
Keywords: Gut virome; Intestinal Bowel Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Ulcerative Colitis (UC): Patients with ulcerative colitis undergoing endoscopy and biopsies-collection according to the standard of care. First diagnosis for UC, treatment naive patients (≥18 and <40 years), with no previously documented gastrointestinal infections. Furthermore, clinical and endoscopic evaluation (Mayo score≥2).
  Interventions: Procedure: Additional biopsies collection
- Crohn's Disease (CD): Patients with Crohn's disease undergoing endoscopy and biopsies-collection according to the standard of care. First diagnosis for CD, treatment naive patients (≥18 and <40 years), with no previously documented gastrointestinal infections. Furthermore, clinical and endoscopic evaluation (Harvey-Bradshaw score≥5 and overall Simplified Endoscopic Score (SES-CD)> 2).
  Interventions: Procedure: Additional biopsies collection
- No UC and CD: Subjects undergoing endoscopy and biopsies-collection according to the standard of care (≥18 and <40 years) (for example patients in screening for colorectal cancer disease). Subjects not affected by UC or CD according to the previously reported clinical and endoscopic evaluation criteria.
  Interventions: Procedure: Additional biopsies collection

INTERVENTIONS:
Procedure: Additional biopsies collection — We will recruit only subjects (UC, CD and NO-UC/CD) scheduled for the endoscopy and biopsies-collection according to the usual clinical practice. During the endoscopy we will collect 6 additional biopsies.

SUMMARY:
Alterations in the composition of the intestinal microbiota (dysbiosis) are well known involved in the pathogenesis of gastrointestinal disorders, such as inflammatory bowel disease (IBD), which includes ulcerative colitis (UC) and Crohn's disease (CD). While bacteria have always gotten the most attention in gastrointestinal disorders, the viral component of the human gut microbiome, called the "gut virome", is underestimated. In addition to bacteriophages, the gut virome also harbors viruses that infect eukaryotic cells, capable of transferring their information directly to host cells, and associated with the pathogenesis of both UC and CD.

Although a substantial number of studies have described the viral composition of gut microbiota in human feces, it is necessary to define the entire eukaryotic virome which colonizes the intestinal mucosa of patients with inflammatory bowel disease and which intestinal cell population is most affected. Therefore, this study aims at a comprehensive metagenomic analysis on single cells of the intestinal mucosa from a large cohort of treatment-naïve young patients with IBD at their first diagnosis to find out which cells are affected by eukaryotic viruses in the early stages of the onset of IBD and how it can affect the immune response of the mucosa, eventually leading to chronic intestinal inflammation.

DETAILED DESCRIPTION:
The human intestine is progressively colonized after birth by several microbial strains that change during lifespan according to anatomical, dietary and nutritional statuses. Alterations in the gut microbiota composition (dysbiosis) are well-recognized contributors to the pathogenesis of gastrointestinal disorders, such as inflammatory bowel disease (IBD), including ulcerative colitis (UC) and Crohn's disease (CD). In fact, bacteria, fungi, archaea, and viruses, all populating the human intestine, were found to control gut homeostasis, with a continuous pathogen-host interplay that results in both local (mucosal and luminal) and systemic (metabolic and nutritional) effects.

Although bacteria have always gained the greatest attention in gastrointestinal disorders, the viral component of the human gut microbiome, termed the "gut virome", is understudied. The viral community of the microbiota is mainly composed of prokaryotic-infecting viruses (bacteriophages), thus rendering the gut a dynamic community structure, characterized by continuous "predator-prey interactions" that cause either horizontal gene transfer (viruses to bacteria) or modification in the bacterial composition of the microbiota, impacting on both health and disease.

Besides bacteriophages, the gut virome hosts also DNA- and RNA-based eukaryotic-targeting viruses able to directly transfer their genetic information to host cells, and demonstrated to be associated with the pathogenesis of both UC and CD. Furthermore, eukaryotic viruses have been shown to contribute to intestinal dysbiosis in mice carrying mutations in the IBD-associated Il10 or Atg16L1 genes, suggesting that the gut virome might cooperate with genetic factors, ultimately leading to chronic intestinal inflammation.

Variations in gut virome composition have been shown to occur also in pathogenic conditions. In fact, by targeted deep-sequencing analysis of stools from patients with CD and UC, Norman and colleagues demonstrated not only that the virome composition was disease- and cohort-specific, but also that its variations contributed to intestinal dysbiosis. However, this study is incomplete, since it exploits metagenomic analysis of DNA sequences only, thus ignoring RNA viruses, such as Norovirus and Astrovirus, previously suggested as potential precipitators or triggers of intestinal inflammation.

Therefore, although a consistent number of studies described the viral composition of the intestinal microbiota in human stools, mainly focusing on bacteriophages, the whole eukaryotic virome that colonizes intestinal mucosa of IBD patients and which intestinal cell population is mainly affected still need to be defined. So far, the occurrence of gut viral infections has been evaluated only in cohorts of IBD patients with long-lasting chronic intestinal inflammation. However, in these studies, either immunosuppressants or disease-induced stressing conditions may have led to the activation of latent viral infections such as those from Hepatitis B and C (HBV and HCV), Cytomegalovirus (CMV) and Epstein-Bar virus (EBV). For example, a recent metagenomic analysis on colonic mucosae revealed Herpesviridae as the most enriched viral community in IBD patients. Nonetheless, since in these works most of the enrolled patients were under pharmacological treatments and not early diagnosed, the identification of any putative viral entity responsible for the onset of IBD might not have been accurate.

The role of viruses in causing and sustaining diseases has been confirmed for tumors so that viral infections are known to be responsible for about 20% of the global cancer burden. Similar to gastrointestinal disorders, also in tumors bacteria and viruses not only influence each other leading to a prevalence or reduction of specific microbe species, but they also synergistically impact on host's immune response.

Overall, these pieces of evidence shed light on novel insights on the role of gut virome in triggering an immune response, by likely conferring to the host a "virus-specific genetic predisposition" (virotype) susceptible to IBD development. Therefore, such aspect of IBD pathogenesis strongly warrants further investigations.

This proposal aims at a comprehensive single-cell population metagenomic analysis of gut mucosae from a large cohort of treatment-naïve young patients with IBD at their first diagnosis to discover which cells are affected by eukaryotic viruses in the initial phases of IBD onset and how they can influence the whole mucosa's immune response, eventually leading to the chronic intestinal inflammation. Results obtained will represent a significant step forward with respect to the previous studies because they will shed light on novel molecular mechanisms through which eukaryotic viruses may lead to gut chronic inflammation, paving the way to the development of novel biomarkers for the diagnosis and drugs for the treatment of IBD.

ELIGIBILITY:
Inclusion Criteria:

SUBJECTS AFFECTED BY UC OR CD:

* subjects undergoing endoscopy and biopsies-collection according to the standard of care first diagnosis for UC or CD, treatment naive patients (≥18 and <40 years)
* no previously documented gastrointestinal infections

Furthermore, for subjects with UC:

- clinical and endoscopic evaluation (Mayo score≥2)

Furthermore, for subjects with CD:

- clinical and endoscopic evaluation (Harvey-Bradshaw score≥5 and overall Simplified Endoscopic Score (SES-CD)> 2)

SUBJECTS NOT AFFECTED BY UC OR CD (CONTROL GROUP):

* subjects undergoing endoscopy and biopsies-collection according to the standard of care (≥18 and <40 years) (for example patients in screening for colorectal cancer disease.)
* subjects not affected by UC or CD according to the previously reported clinical and endoscopic evaluation criteria

All patients will be asked to sign the written informed consent.

Exclusion Criteria:

SUBJECTS AFFECTED BY UC OR CD:

* subjects with UC or CD who do not respect the clinical and endoscopic evaluation criteria previously described
* subjects with UC or CD who respect the clinical and endoscopic evaluation criteria BUT previously treated with/undergoing anti-inflammatory and/or immunosuppressive drugs

SUBJECTS NOT AFFECTED BY UC OR CD (CONTROL GROUP):

- subjects undergoing anti-inflammatory and/or immunosuppressive treatments for other diseases not related to UC or CD

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: We will recruit adult naïve patients with colitic CD or UC at their first diagnosis, ≥18 and <40 years and without any previously documented gastrointestinal infections in collaboration with the Gastroenterology and Digestive Endoscopy unit (IRCSS Ospedale San Raffaele).
  CD and UC diagnosis will be determined by clinical and endoscopic scores (described in inclusion criteria). Control data will come from the same intestinal areas of age-matched no-UC/CD subjects undergoing endoscopic surveillance for not IBD-related conditions according to the standard of care.
  The participation is voluntary and the patient is allowed to refuse further participation in the protocol whenever he/she wants.
Sampling Method: Probability Sample
Enrollment: 69 (Estimated)
Dates: Start 2023-02-07 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Characterization of the gut virome | 13 months
  To collect and characterize scpRNAseq-transcriptomes derived from intestinal mucosa of early-diagnosed, treatment naïve young IBD patients

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No